CLINICAL TRIAL: NCT07028203
Title: Evaluation of the Safety and Efficacy of the BTL-785 Device for Non-invasive Rejuvenation of the Periorbital Area and Lower Eyelid
Brief Title: Non-invasive Rejuvenation of the Periorbital Area and Lower Eyelid
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS1800
Record Dates: First submitted 2025-06-09; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Periorbital Wrinkles; Periorbital Area; Under-eyes Dark Circles; Crows Feet
Keywords: under-eye bags; dark circles; periorbital; crows feet
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with BTL-785 with the applicator BTL-785-7-11 (Experimental): The treatment administration phase will consist of four treatment visits.
  Interventions: Device: Treatment with BTL-785 with the applicator BTL-785-7-11

INTERVENTIONS:
Device: Treatment with BTL-785 with the applicator BTL-785-7-11 — The treatment administration phase will consist of four (n=4) treatments, delivered 2 -14 days apart. The applicator will be placed outside the orbital rim, on the subject's inferior orbital portion of the orbicularis oculi muscles and lateral canthal edge-temporal area. Therapy time is set to 20 minutes.

SUMMARY:
The goal of this clinical trial is to determine the BTL-785-7-11 applicator effectiveness for an under-eye appearance improvement by evaluation of the periorbital area in healthy adult volunteers. The main question it aims to answer is:

Whether the BTL-785-7-11 applicator is able to improve the periorbital area post-treatment, as assessed by the analysis of 3D photographs.

Participants will complete four treatments and two follow-up visits.

DETAILED DESCRIPTION:
The study will evaluate the clinical efficacy and safety of the BTL-785 device with applicator BTL-785-7-11 for periorbital area rejuvenation.

The study has a prospective, multicenter, open-label, and one-arm design.

Subjects will be required to complete four (n=4) treatment visits and two (n=2) follow-up visits.

At the baseline visit, inclusion and exclusion criteria will be verified upon obtaining informed consent from the patient. Digital 2D and 3D photographs of the treatment area will be taken.

The treatment administration phase will consist of four (n=4) treatments, delivered 2 -14 days apart. The applicator will be placed outside the orbital rim, on the subject's inferior orbital portion of the orbicularis oculi muscles and lateral canthal edge-temporal area. Therapy time is set to 20 minutes. At the last therapy visit, the subject's digital 2D and 3D photographs of the treatment area will be collected. In addition, subjects will receive therapy comfort and subject satisfaction questionnaires to fill in.

During the 1-month and 3-month follow-up visits, the subjects will undergo 2D and 3D photographing of the treatment area, and the subject satisfaction questionnaires will be collected.

Safety measures will include documentation of adverse events (AE), which will be assessed after each procedure and at all follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking aesthetic improvement of the periorbital area
* Subjects should be able to understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible aging signs in the periorbital area (e.g. under-eye bags, periorbital wrinkles) when the face is relaxed as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Lower eyelid malposition (ectropion, entropion, retraction)
* Blepharitis
* Prior lower eyelid fat removal, skin resection, eyelid surgery or orbital trauma in the past 6 months, prior dermatochalasis of lower eyelids surgical treatment in the past 6 months
* Filler injections in the treatment area and midface region within 3 months prior to the study participation
* Neuromodulator treatment in the periorbital area within 3 months prior to the study participation
* Tattoo(s) and/or permanent make-up in the intended treatment area
* Prior usage within 30 days before the screening or planned usage during the study of retinol, or any medication that can cause dermal hypersensitivity
* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin-related autoimmune diseases
* Radiation therapy and chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants near treatment area or neutral electrode
* Permanent implant near the area to be treated
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Current condition or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of malignant cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Electroanalgesia without exact diagnosis of pain etiology
* Tuberculosis
* Hepatitis
* Febrile conditions
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Sensitive disorders in the treatment area
* Varicose veins, pronounced edemas
* Skin dermabrasion, skin resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Application in the area of chest, heart, carotid sinus, mouth (i.e. over the lips and in the near proximity) or over the eyes (i.e. over the eyeballs and eyelids)
* Serious psychopathological disorders (such as schizophrenia)
* Neurological disorders (such as multiple cerebrospinal sclerosis, epilepsy)
* Blood vessels and lymphatic vessels inflammation
* Scarring in the treatment area

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-11-09 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Periorbital area improvement assessment | baseline to 3 months post-treatment
  The evaluation of the periorbital area improvement comparing pre-treatment, the last therapy visit, and both 1-month and 3-month follow-up visits will be based on the analysis of 3D photographs.

SECONDARY OUTCOMES:
Assessment of changes in the visual appearance, according to the Global Aesthetic Improvement Scale | baseline to 3 months post-treatment
  The assessment of changes in the visual appearance will be based on the evaluation of the 2D photographs, according to the Global Aesthetic Improvement Scale (GAIS); the ranking is based on the 5-point scale (ranging from -1 to 3), higher score means a more improved appearance.
Assessment of changes in the visual appearance, according to the Fitzpatrick Wrinkle and Elastosis Scale | baseline to 3 months post-treatment
  The assessment of changes in the visual appearance will be based on the evaluation of the 2D photographs, according to the Fitzpatrick Wrinkle and Elastosis Scale (FWES); the ranking is based on the 10-point scale (ranging from 0 to 9), higher score means a more severe aesthetic condition being evaluated.
Assessment of changes in the visual appearance, according to the Crow's Feet Grading Scale | baseline to 3 months post-treatment
  The assessment of changes in the visual appearance will be based on the evaluation of the 2D photographs, according to the Crow's Feet Grading Scale (CFGS); the ranking is based on the 5-point scale (ranging from 0 to 4), higher score means a more severe crow's feet.
Subject satisfaction as assessed by Subject Satisfaction Questionnaire | baseline to 3 months post-treatment
  Subject Satisfaction evaluation based on the Subject Satisfaction Questionnaire; the ranking is based on the 5-point Likert scale (1-5), higher score means higher satisfaction.
Comfort as assessed by Therapy Comfort Questionnaire | from the first to the last treatment session, assessed up to 56 days
  Therapy comfort evaluation through the Therapy Comfort Questionnaire; the ranking is based on the 5-point Likert scale (1-5), higher score means higher comfort, and on the Numerical Analog scale (0-10), higher score means higher pain.
Incidence of Treatment-related Adverse Events | baseline to 3 months post-treatment
  Assessment of safety by evaluating the side effects and AE occurrence throughout the study.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Laser & Skin Surgery Medical Group, Inc., Sacramento, California
  - Art of Skin MD, Solana Beach, California
  - Gentile Facial Plastic and Aesthetic Laser center, Youngstown, Ohio